CLINICAL TRIAL: NCT01153685
Title: Immunogenicity and Safety Study of GSK Biologicals' (GSK1536489A) Trivalent Split Virion Influenza Vaccine Fluviral® (2010 - 2011 Season) in Adults Aged 18 to 60 Years and Over 60 Years.
Brief Title: Immunogenicity & Safety Study of Fluviral® (2010 - 2011 Season) in Adults Aged 18 to 60 Years and Over 60 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110628
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Fluviral®Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral A Group (Experimental): Subjects aged between 18 and 60 years who received one dose of Fluviral vaccine at Day 0, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluviral®
- Fluviral B Group (Experimental): Subjects over 60 years of age who received one dose of Fluviral vaccine at Day 0, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluviral®

INTERVENTIONS:
Biological: Fluviral® — Intramuscular injection, one dose

SUMMARY:
This study is designed to test the safety and immunogenicity of Fluviral® (2010 - 2011 Season) in adults aged 18 to 60 years and over 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject
* Male and female adults, 18 to 60 years of age and over 60 years of age.
* Satisfactory baseline medical assessment by history and physical examination
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Participation in previous year's (2009) Fluviral registration study
* Administration of any influenza vaccine within 6 months preceding the study start (35 or more subjects in the >60 year old age stratum will be recruited from among those who did NOT receive any inactivated influenza vaccine in 2009-2010 season, i.e. seasonal TIV or pandemic H1N1v).
* Administration of any other vaccine(s) within 30 days prior to study enrollment or during the study period. Subjects who receive such treatment after enrollment will be followed per protocol and included in the safety analysis, but excluded from the according-to-protocol cohort.
* Clinically or virologically confirmed influenza infection within 1 year preceding the study start.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. oral temperature <38.0°C.
* Significant acute or chronic, uncontrolled medical or psychiatric illness. "Uncontrolled" is defined as:

  * Requiring institution of new medical or surgical treatment within one (1) month prior to study enrollment, or
  * Requiring the re-institution of a previously discontinued medication or medical treatment within one month prior to study enrollment, or
  * Requiring a change in medication dosage in the one month prior to study enrollment due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  * Hospitalization or an event fulfilling the definition of a SAE within one month prior to study enrollment.
* Any confirmed or suspected immunosuppressive condition including:

  * History of human immunodeficiency virus (HIV) infection,
  * Cancer or treatment for cancer, within 3 years of study enrollment. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* History of renal impairment.
* History of hepatic dysfunction due to hepatitis B, C or toxins including alcohol.
* Complicated insulin-dependent diabetes mellitus.
* Unstable cardiopulmonary disease requiring chronic medical therapy or associated with functional impairment.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* Receipt of systemic glucocorticoids (prednisone >= 20 mg/day for more than 14 consecutive days) within 1 month of study enrollment, or any cytotoxic or immunosuppressive drugs within six months of study enrollment. Inhaled and topical steroids are allowed.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* History of chronic alcohol consumption and/or drug abuse.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin. Persons receiving prophylactic antiplatelet medications, e.g. low-dose aspirin, and without a clinically-apparent bleeding tendency are eligible.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of Fluviral (egg protein, thimerosal) and/or a history of anaphylactic type reaction to consumption of eggs, and/or reactions to products containing mercury (such as thimerosal).
* A history of severe adverse reaction to a previous influenza vaccination.
* Pregnant and/or lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07-09; Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jain VK, Chandrasekaran V, Wang L, Li P, Liu A, Innis BL. A historically-controlled Phase III study in adults to characterize the acceptability of a process change for manufacturing inactivated quadrivalent influenza vaccine. BMC Infect Dis. 2014 Mar 10;14:133. doi: 10.1186/1471-2334-14-133. PMID 24606983
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluviral A Group | Fluviral B Group
Started | 50 | 70
Completed | 50 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral A Group | Fluviral B Group | Total
Number analyzed (Participants) | 50 | 70 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (13.72) | 66.6 (4.73) | 50.7 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 17 | 31 | 48

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Haemagglutination Inhibition (HI) Antibodies Against Fluviral Vaccine Strains.
Description: The Fluviral vaccine strains were A/California (H1N1), A/Victoria (H3N2) and B/Brisbane
Time Frame: At Day 0 before vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Titer
  A/California (H1N1) | 39.2 [24.0 to 63.8] | 15.2 [11.1 to 21.0]
  A/Victoria (H3N2) | 14.1 [10.1 to 19.8] | 13.0 [9.8 to 17.3]
  B/Brisbane | 22.7 [15.2 to 34.0] | 28.0 [21.5 to 36.5]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Haemagglutination Inhibition (HI) Antibodies Against Fluviral Vaccine Strains.
Description: The Fluviral vaccine strains were A/California (H1N1), A/Victoria (H3N2) and B/Brisbane
Time Frame: At Day 21 after vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Titer
  A/California (H1N1) | 390.1 [293.8 to 518.1] | 142.1 [105.1 to 192.0]
  A/Victoria (H3N2) | 185.6 [140.9 to 244.5] | 183.7 [139.6 to 241.8]
  B/Brisbane | 260.6 [184.6 to 368.0] | 248.6 [185.9 to 332.3]

3. Primary Outcome: Number of Seroprotected Subjects for Antibodies Against Fluviral Vaccine Strains.
Description: A Seroprotected subject was defined as a subject with a serum haemagglutination inhibition (HI) antibody titer greater than or equal to 1:40.
Time Frame: At Day 0 before vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Subjects
  A/California (H1N1) | 29 | 22
  A/Victoria (H3N2) | 15 | 17
  B/Brisbane | 21 | 35

4. Primary Outcome: Number of Seroprotected Subjects for Antibodies Against Fluviral Vaccine Strains.
Description: as for outcome 3
Time Frame: At Day 21 after vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Subjects
  A/California (H1N1) | 49 | 62
  A/Victoria (H3N2) | 48 | 65
  B/Brisbane | 47 | 69

5. Primary Outcome: Number of Seroconverted Subjects for Antibodies Against Fluviral Vaccine Strains.
Description: A subject seroconverted for haemagglutination inhibition (HI) antibodies was defined as a subject with either a prevaccination (Day 0) HI antibody titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a prevaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 21 after vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Subjects
  A/California (H1N1) | 35 | 50
  A/Victoria (H3N2) | 41 | 57
  B/Brisbane | 33 | 51

6. Primary Outcome: Seroconversion Factor for Antibodies Against Fluviral Vaccine Strains.
Description: Seroconversion Factor (SCF) is defined as the fold increase in serum HI antibody GMTs post-vaccination (Day 21) compared to prevaccination (Day 0).
Time Frame: At Day 21 after vaccination
Population: The analyses were based on the According-To-Protocol (ATP) cohort for immunogenicity.
Measure: Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 49 | 70
Fold increase
  A/California (H1N1) | 10.0 [6.3 to 15.7] | 9.3 [6.8 to 12.8]
  A/Victoria (H3N2) | 13.1 [9.3 to 18.5] | 14.1 [10.2 to 19.5]
  B/Brisbane | 11.5 [7.0 to 18.7] | 8.9 [6.3 to 12.4]

7. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms After Administration of Fluviral.
Description: Solicited local symptoms assessed were pain, redness and swelling at the injection site. Solicited general symptoms assessed were bronchospasm, chills, cough, fatigue, headache, joint pain at other location, muscle aches, red eyes, sore throat, swelling of the face and temperature (defined as orally temperature equal or above 38.0 degrees Celcius)
Time Frame: During a 4-days (Day 0-3) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated Cohort on subjects with available results.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 50 | 69
Subjects
  Pain | 41 | 18
  Redness | 0 | 0
  Swelling | 2 | 1
  Bronchospasm | 0 | 3
  Chills | 2 | 0
  Cough | 2 | 0
  Fatigue | 15 | 7
  Headache | 13 | 6
  Joint pain at other location | 6 | 3
  Muscle aches | 17 | 6
  Red eyes | 4 | 1
  Sore throat | 8 | 2
  Swelling of the face | 1 | 0
  Temperature | 1 | 1

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse events (AE) covers any AE reported in addition to those solicited during the clinical study and any solicited symptoms with onset outside the specified period of follow-up for solicited symptoms.
  Any = occurrence of any adverse event regardless of intensity grade or relationship to vaccination.
  Grade 3 = an unsolicited AE that prevented normal everyday activity. Related = event assessed by the investigator as causally related to the vaccination.
Time Frame: Within the 21-day post-vaccination period
Population: The analysis was performed on the Tota Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 50 | 70
Subjects
  Any | 16 | 17
  Grade 3 | 1 | 0
  Related | 8 | 3

9. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 21-day post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 50 | 70
Subjects
  Headache | 1 | 3
  Nausea | 3 | 1
  Diarrhoea | 3 | 0
  Dizziness | 1 | 2
  Abdominal pain | 2 | 0
  Cough | 0 | 2
  Back pain | 0 | 1
  Breast pain | 0 | 1
  Conjunctivitis | 1 | 0
  Contusion | 1 | 0
  Crohn's disease | 1 | 0
  Depression | 1 | 0
  Dysmenorrhoea | 1 | 0
  Ear pain | 1 | 0
  Epididymitis | 0 | 1
  Fatigue | 1 | 0
  Folliculitis | 1 | 0
  Gingival pain | 1 | 0
  Injection site haematoma | 1 | 0
  Injection site pain | 1 | 0
  Injection site paraesthesia | 1 | 0
  Insomnia | 1 | 0
  Localized infection | 0 | 1
  Menorrhagia | 1 | 0
  Metrorrhagia | 1 | 0
  Mouth ulceration | 1 | 0
  Musculoskeletal chest pain | 1 | 0
  Musculoskeletal pain | 0 | 1
  Nasopharyngitis | 0 | 1
  Ocular hyperaemia | 0 | 1
  Pain | 0 | 1
  Procedural pain | 0 | 1
  Renal colic | 1 | 0
  Sedation | 1 | 0
  Sinus headache | 0 | 1
  Sleep apnoea syndrome | 0 | 1
  Tooth fracture | 0 | 1
  Urinary tract infection | 0 | 1
  Vomiting | 1 | 0

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period
Population: The analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | Fluviral A Group | Fluviral B Group
Number analyzed (Participants) | 50 | 70
Subjects | 2 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during a 4-day follow-up period after vaccination. Unsolicited symptoms: during 21 days following the vaccination (Day 0-21). Serious adverse events: during the entire study period (21 days)
Arm/Group | Fluviral A Group | Fluviral B Group
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/70
Other Adverse Events (participants affected / at risk) | 45/50 | 30/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral A Group (N=50) | Fluviral B Group (N=70)
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluviral A Group (N=50) | Fluviral B Group (N=70)
Pain (General disorders) | 41 | 18/69
Fatigue (General disorders) | 15 | 7/69
Headache (Nervous system disorders) | 13 | 6/69
Joint pain at other location (General disorders) | 6 | 3/69
Muscle aches (Musculoskeletal and connective tissue disorders) | 17 | 6/69
Red eyes (Eye disorders) | 4 | 1/69
Sore throat (Infections and infestations) | 8 | 2/69
Nausea (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.